CLINICAL TRIAL: NCT06752278
Title: Efficacy of Pilocarpine As a Secretagogue Versus Artificial Tears for the Treatment of Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab Tharwat, Prinicipal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pilocarpine and Dry Eye
Record Dates: First submitted 2024-12-27; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Pilocarpine; Lubricant Eye Drops

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pilocarpine group (Active Comparator)
  Interventions: Drug: Pilocarpine
- artificial tears group (Active Comparator)
  Interventions: Drug: artificial tears

INTERVENTIONS:
Drug: Pilocarpine — Pilocarpine is a muscarinic agonist
  Arms: pilocarpine group
Drug: artificial tears — artificial tears used for the treatment of Dry eye
  Arms: artificial tears group

SUMMARY:
Management approaches for dry eye disease (DED) typically start with low-risk, easily accessible, patient-applied therapies like artificial tears for early-stage disease. As the condition worsens, treatment progresses to more advanced therapies for severe forms of DED. This study aims to compare the effectiveness and safety of pilocarpine as a secretagogue versus artificial tears in the treatment of dry eye disease. Our goal is to provide reliable, high-quality evidence regarding the efficacy of secretagogues, thereby contributing to the development of recommendations that aid clinicians in their decision-making process

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with DED

Exclusion Criteria:

* Previous Occular surgery.
* Refuse to particupate.
* Patients with sjogren syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index | At the baseline and after 6 weeks
tear film break-up time | At the baseline and after 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar university, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided